CLINICAL TRIAL: NCT02596906
Title: Brain and Cognitive Changes After Reasoning Training in Individuals With Cognitive Complaints
Brief Title: Brain and Cognitive Changes After Reasoning Training in Individuals With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sandra Chapman, PhD, Director, Center for BrainHealth, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBH-MCI-tDCS
Record Dates: First submitted 2015-10-30; First posted 2015-11-04 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- tDCS+Training (Experimental): This group will receive 20 minutes of tDCS, 8x over four weeks immediately followed by reasoning training 8x over four weeks
  Interventions: Device: tDCS
- Sham tDCS+training (Sham Comparator): This group will receive 20 minutes of "sham" tDCS, 8x over four weeks immediately followed by reasoning training 8x over four weeks.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — Prior to the reasoning training, participants will undergo tDCS. Participants will receive 20 minutes of tDCS using 2mA or less targeting the inferior frontal gyrus prior to each of their 8 reasoning training sessions for a total of 160 total combined minutes. This time does not include set up time which should take no more than 5 minutes. A brief engaging film is shown to participants during the 20 minute session.
  Arms: tDCS+Training
Device: Sham tDCS — For the sham tDCS group, the device will be turned off after 30s. The only reported sensations from tDCS is an itching or a tingling when the device turns on but disappears quickly. Thus, those receiving sham tDCS will be unaware that the device has turned off, and will experience an initial tingling similar to that received in the tDCS group.
  Arms: Sham tDCS+training

SUMMARY:
Individuals aged 55 and older may experience negative effects of cognitive decline. The proposed research seeks to evaluate the benefits of different types of interventions: reasoning training following transcranial direct current stimulation (tDCS) and reasoning training following sham transcranial direct current stimulation (tDCS) on frontal- lobe mediated cognitive measures of executive control in adults with memory complaints, in the absence of dementia.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of reasoning training on individuals with complaints of changes in memory or thinking in the absence of dementia, when combined with transcranial current stimulation (tDCS). The reasoning training being studied is a strategy based program where individuals are taught strategies designed to engage the frontal lobes. Participants will randomly be placed into one of two groups (1) reasoning training following transcranial current stimulation (tDCS) as compared to (2) reasoning training following sham tDCS. The study will be done with adults between the ages of 50 and 80 with consistent memory complaints or lower baseline performance on memory measures. The primary hypothesis is that individuals receiving tDCS prior to brain training will have a stronger response to brain training than those in the sham tDCS group. Response to training will be measured by improved cognitive function and neural changes as measured by neuropsychological testing, MRI, and EEG. MRI will be used to evaluate the impact of reasoning training on brain blood flow, structure and function, and to measure changes in brain energy metabolism and electroencephalogram (EEG) to evaluate intervention outcomes. The reasoning training program will be conducted in small groups at the Center for BrainHealth.

ELIGIBILITY:
Inclusion Criteria:

* Safely have an MRI
* Cognitive complaints in the absence of dementia
* Participate in tasks involving motor abilities such as use of at least one arm and hand
* Read, speak, and comprehend English
* 50-80 years of age
* Comprehend simple instructions, perform tasks, and take part in intervention

Exclusion Criteria:

* Not proficient in reading, comprehending, or speaking English
* Individuals who have any significant health, neurological, or psychiatric illness, or history of substance abuse
* Individuals with any MR contraindications (i.e., non-removable metal within/on the body)
* Individuals taking medications which are contraindicatory for the tDCS procedure
* Individuals who are left-handed
* Not proficient in reading,comprehending, and speaking English
* Females who are not post-menopausal
* Pre-existing cerebral palsy, autism, epilepsy, schizophrenia, pervasive developmental disorder, thyroid diseases, diabetes, claustrophobia, non-correctable vision problems, major depression, psychosis, active behavioral disorder, or uncontrolled epilepsy.
* Women who are pregnant

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Chapman, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- UTD Center for BrainHealth, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu WY, Ku Y, Zanto TP, Gazzaley A. Effects of noninvasive brain stimulation on cognitive function in healthy aging and Alzheimer's disease: a systematic review and meta-analysis. Neurobiol Aging. 2015 Aug;36(8):2348-59. doi: 10.1016/j.neurobiolaging.2015.04.016. Epub 2015 May 1. PMID 26022770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 participants consented for the study of which 15 were included in the final analysis.
Pre-assignment Details: 331 participants were screened for eligibility criteria, of which 52 participants were eligible for the study. Of the 52, a total of 30 participants dropped out due to time constraints, inability to complete the scans and/or after recommendation by the neurologist who questioned if they truly met eligibility criteria.
Period: Overall Study
Arm/Group | tDCS+Training | Sham tDCS+Training
Started (The units assigned is indeed the participants) | 12 | 10
Completed (3-month follow-up) | 8 | 7
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Population: Individuals in this study had memory complaints as supported by objective cognitive testing but were functionally independent. A neurologist confirmed the diagnosis of mild cognitive impairment based on objective cognitive testing.
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS+Training | Sham tDCS+Training | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Overall, the number of participants completed the cognitive training and tDCS stimulation protocol is 32 of which only 22 participant data were useable. The reason for attrition is due to either noncompliance of training or unable to use the MRI data due to movement.
  years | 64.17 (6.93) | 63.30 (7.38) | 63.91 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Overall, the number of participants completed the cognitive training and tDCS stimulation protocol is 32 of which only 22 participant data were useable. The reason for attrition is due to either noncompliance of training or unable to use the MRI data due to movement.
  Participants
    Female | 5 | 6 | 11
    Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in California Verbal Learning Task Score
Description: To examine short-term and long-term effects of treatment on cognition and real-life outcomes. The participant will undergo neuropsychological testing at baseline, post-training (4 weeks), as well as 3-months post-training.
  Scores on the scale range from 0 to 16 on the California Verbal Learning Task. Higher the values are better their memory.
Time Frame: Baseline to 4 weeks and 3 months post-training
Population: 22 participants consented to the study of which 15 participants were in the final analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS+Training | Sham tDCS+Training
Number analyzed (Participants) | 8 | 7
score on a scale
  Baseline to 4 weeks | 3.04 (1.22) | 5.17 (2.22)
  Baseline to 3-month follow-up | 4.22 (1.45) | 7.04 (1.44)

2. Secondary Outcome: Regional Brain Blood Flow Change Immediately After 1 Month of Cognitive Training and tDCS Brain Stimulation
Description: Non-invasive estimation of rCBF by perfusion maps using pseudo-continuous arterial spin labeling (pCASL) MRI. rCBF is quantified as mL/min/100g tissue.
Time Frame: Two longitudinal measurements at baseline and 1-month
Population: Participants between ages 50-80 years had a diagnosis of mild cognitive impairment (MCI)based on Petersen's or Alzheimer's Disease Neuroimaging Initiative (ADNI) criteria from the Dallas-Fort worth community.
Measure: Mean (95% Confidence Interval); unit: ml/min/100g tissue scaled by whole brain
Arm/Group | tDCS+Training | Sham tDCS+Training
Number analyzed (Participants) | 8 | 7
ml/min/100g tissue scaled by whole brain | 0.19 [0.04 to 0.34] | -0.12 [-0.27 to 0.03]

ADVERSE EVENTS:
Time Frame: Baseline to 4 months
Description: Two participants had adverse events in the study: 1 participant had a minor burn from the tDCS and a 2nd participant became dizzy and vomited at the scanner.
Arm/Group | tDCS+Training | Sham tDCS+Training
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 2/8 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 0.167% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS+Training (N=8) | Sham tDCS+Training (N=7)
Baseline at 1pm on June 26th 2017 for 15 minutes (Gastrointestinal disorders) | 1 (1) | 0 (0) — The participant experienced dizziness in the 7T scanner, which persisted past the initial few minutes of the scan.
Baseline on February 26th 2017 for 1week on March 2nd 2017 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — One subject observed a burn on the right deltoid the site of tDCS stimulation electrode. The scar subsided in 1 week

LIMITATIONS AND CAVEATS:
Participant enrollment was limited due to constraints on time and funding sources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT02596906/Prot_SAP_001.pdf